CLINICAL TRIAL: NCT00288704
Title: IL1T-AI-0505: A Multi-center, Double-Blind, Placebo-Controlled Study of the Safety, Tolerability, & Efficacy of Rilonacept in Subjects With Cryopyrin-Associated Periodic Syndromes (CAPS) Using Parallel Group & Randomized Withdrawal Designs
Brief Title: Rilonacept for Treatment of Cryopyrin-Associated Periodic Syndromes (CAPS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IL1T-AI-0505
Record Dates: First submitted 2006-02-06; First posted 2006-02-08 (Estimated); Results first posted 2009-11-13 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Familial Cold Autoinflammatory Syndrome (FCAS); Familial Cold Urticaria; Muckle-Wells Syndrome (MWS); Genetic Diseases, Inborn
Keywords: Familial Cold Autoinflammatory Syndrome (FCAS); Muckle-Wells Syndrome (MWS); CIAS1; NLRP-3; PYPAF1; Cryopyrin; CAPS; Interleukin-1
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes; Genetic Diseases, Inborn | interventions — rilonacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Some subjects were treated with Placebo in the Study. This occurred (if subject randomized to Placebo) either during the first 6 weeks of the study or during the randomized withdrawal (weeks 15-24).
  Interventions: Drug: Placebo
- rilonacept 160 mg (Active Comparator): If randomized to rilonacept, subjects received this treatment during the first 6 weeks of the study or during the randomized withdrawal (weeks 15-24). All subjects received rilonacept 160 mg during weeks 6-14 (between Parts A and B).
  Study drug is administered as a 2.0 mL subcutaneous injection once a week. At baseline (week 0) subjects receive a loading dose of rilonacept 320 mg.
  Interventions: Drug: rilonacept 160 mg
- Open-Label rilonacept 160 mg (Other): After week 24 (the end of part B), all subjects went into weekly dosing of open label rilonacept 160 mg. During this phase of the study, adolescents aged 7 and above were entered into the study and rilonacept was dosed as 2.2 mg/kg injections, up to 160 mg, per week.
  Study drug is administered as a 2.0 mL subcutaneous injection once a week.
  Interventions: Drug: rilonacept 160 mg

INTERVENTIONS:
Drug: rilonacept 160 mg — Rilonacept was given by subcutaneous injection. It was administered weekly at the dose of 160mg. On Day 1, subjects received two injections of rilonacept (for a total of 320 mg).
  Other Names: Rilonacept
  Arms: rilonacept 160 mg
Drug: Placebo — Subcutaneous injection of Placebo occurred during first 6 weeks of the study or during randomized withdrawal (weeks 15-24). On Day 1, subjects received two placebo injections.
  Arms: Placebo
Drug: rilonacept 160 mg — Rilonacept was given by subcutaneous injection. It was administered weekly at the dose of 160mg. No loading dose was given for subjects who entered directly into the open-label.
  Arms: Open-Label rilonacept 160 mg

SUMMARY:
Inflammatory symptoms of Cryopyrin-Associated Periodic Syndrome (CAPS) are due to mutations in a the NLRP-3 gene (previously known as Cold Induced Autoinflammatory Syndrome-1 or CIAS1). These mutations result in the body's overproduction of interleukin-1 (IL-1), a protein that stimulates the inflammatory process. IL-1 Trap (rilonacept) was designed to bind to the interleukin-1 cytokine and prevent it from binding to its receptors in the body.

DETAILED DESCRIPTION:
Primary Objective:

The primary objective of this study was to assess the effect of rilonacept on the clinical signs and symptoms of Cryopyrin-Associated Periodic Syndrome (CAPS) when used for chronic therapy as evaluated by the subjects themselves over time using a validated patient-reported outcomes tool.

Secondary Objective(s):

The secondary objectives were as follows:

* To determine the safety and tolerability of rilonacept in subjects with CAPS
* To assess the effect of rilonacept on laboratory measures of inflammation such as acute phase reactants

This was a multi-center, two-part, double-blind, placebo-controlled study (Parts A and B) designed to assess the efficacy, safety, and tolerability of weekly subcutaneous (SC) doses of 160 mg of rilonacept in adult subjects with active CAPS. These phases were followed by extended open-label phases. After written informed consent was obtained, subjects who met the protocol eligibility criteria were enrolled at one of 27 study sites in the United States. The study consisted of a 3-week screening period preceding Part A, a 6-week long double-blind, randomized phase of the study. All subjects were then treated with single-blind rilonacept for 9-weeks, followed by a subsequent 9-week, double-blind, withdrawal phase during which subjects were re-randomized to either rilonacept or placebo. Subjects then continued treatment in a 24-week open-label extension phase (OLE) and a further 112-week long-term open-label extension (LTOLE), during which all subjects received rilonacept and a 6-week post-treatment follow-up period. Amendments 4 and 6 allowed eligible adult and pediatric subjects aged 7 and above to enroll directly into the open-label phases of the trial.

For reporting purposes, the 24-week OLE and the 112-week LTOLE was considered one Open Label Extension (OLE) phase. This occurred after the 24-week double blind (Parts A and B ) phase. In other words, OLE Week 1 corresponded to the week 25 in the study.

OLE Week 72 was the final timepoint where efficacy was measured. Safety continued after that timepoint until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Double-blind phases: adults age 18 and above; Open-label extension: Adults and children aged 7 years and older.
* Was diagnosed with Familial Cold Auto-inflammatory Syndrome (FCAS) or Muckle-Wells Syndrome (MWS) based upon clinical signs and symptoms
* Had documented mutation in NLRP-3 (Cold Induced Autoinflammatory Syndrome-1 or CIAS1) in subject or relative, and willingness to have a confirmatory genetic (Deoxyribonucleic acid or DNA) test (cheek swab).
* Was able to understand and comply with study procedures and was able to provide informed consent
* If female, was not currently pregnant and was willing to use contraception during the study

Exclusion Criteria:

* Had evidence of untreated tuberculosis or other conditions/therapies that made the subject inappropriate for this study.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2005-12; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Evans, PharmD., Study Director — Regeneron Pharmaceuticals
Locations (24):
- United States (24):
  - Little Rock, Arkansas
  - Palm Desert, California
  - Upland, California
  - Jacksonville, Florida
  - Stuart, Florida
  - Atlanta, Georgia
  - Columbus, Georgia
  - Aurora, Illinois
  - Louisville, Kentucky
  - Shreveport, Louisiana
  - Chesterfield, Michigan
  - St Louis, Missouri
  - New York, New York
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Duncansville, Pennsylvania
  - Columbia, South Carolina
  - Greer, South Carolina
  - Chattanooga, Tennessee
  - Dallas, Texas
  - Waco, Texas
  - Cedar City, Utah
  - Forest, Virginia
  - Lakewood, Washington

REFERENCES:
- [Derived] Hoffman HM, Throne ML, Amar NJ, Cartwright RC, Kivitz AJ, Soo Y, Weinstein SP. Long-term efficacy and safety profile of rilonacept in the treatment of cryopryin-associated periodic syndromes: results of a 72-week open-label extension study. Clin Ther. 2012 Oct;34(10):2091-103. doi: 10.1016/j.clinthera.2012.09.009. Epub 2012 Sep 29. PMID 23031624
- [Derived] Hoffman HM, Throne ML, Amar NJ, Sebai M, Kivitz AJ, Kavanaugh A, Weinstein SP, Belomestnov P, Yancopoulos GD, Stahl N, Mellis SJ. Efficacy and safety of rilonacept (interleukin-1 Trap) in patients with cryopyrin-associated periodic syndromes: results from two sequential placebo-controlled studies. Arthritis Rheum. 2008 Aug;58(8):2443-52. doi: 10.1002/art.23687. PMID 18668535
- See also: click here for more information on rilonacept — http://www.ncbi.nlm.nih.gov/pubmed/18668535?ordinalpos=13&itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_DefaultReportPanel.Pubmed_RVDocSum

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 47 subjects were randomized into Part A. 44 of these subjects continued into the open label extension (OLE). 57 subjects were enrolled directly into the OLE without completing parts A and B of the study. 104 total subjects were in the entire study. 101 were in the OLE.
Pre-assignment Details: The study population included male or female adult subjects (Parts A and B), and adult and pediatric subjects (OLE phase), with confirmed NLRP-3 (Cold Induced Autoinflammatory Syndrome-1 or CIAS1) gene mutation. Only one person per household was enrolled into Parts A and B of the study. However, multiple family members went into the OLE.
Groups:
- Placebo: If assigned, subjects received Placebo during 1) the first 6 weeks of the study (Part A) or 2) during the randomized withdrawal period from weeks 15-24 (Part B). No subject received Placebo during the open-label extension (after week 24). The drug is administered subcutaneously on a weekly basis.
- Rilonacept 160 mg: If assigned, subjects received rilonacept 160 mg during 1) the first 6 weeks of the study (Part A) or 2) during the randomized withdrawal period from weeks 15-24 (Part B). Note: Between weeks 6 and 15 (Parts A and B), all subjects received rilonacept 160 mg.
  Study drug is administered as a 2.0 mL subcutaneous injection once a week. At baseline (week 0) subjects receive a loading dose of rilonacept 320 mg.
- Open-Label Extension (OLE) Rilonacept 160 mg: After week 24 of study, all subjects received weekly injections of rilonacept 160 mg until the end of the study. This was not part of the double blind (Part A) or randomized withdrawal (Part B) portion of the results. Pediatric subjects received rilonacept dosed 2.2 mg/kg weekly up to 160 mg.
  Study drug is administered as a 2.0 mL subcutaneous injection once a week.
Period: Part A, Double Blind, Weeks 1-6
Arm/Group | Placebo | Rilonacept 160 mg | Open-Label Extension (OLE) Rilonacept 160 mg
Started | 24 | 23 | 0 (Subjects enrolled into the open-label phase do not complete this part of the study.)
Completed | 24 | 22 | 0
Not Completed | 0 | 1 | 0
Not completed — Pre-dose Condition | 0 | 1 | 0
Period: Part B, Randomized Withdrawal, Wks 15-24
Arm/Group | Placebo | Rilonacept 160 mg | Open-Label Extension (OLE) Rilonacept 160 mg
Started | 23 (1 subject discontinued during weeks 6-14 due to non-compliance with study drug dosing procedures.) | 22 | 0
Completed | 23 | 21 | 0
Not Completed | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0
Period: Open-Label Extension (OLE) Weeks 24-117
Arm/Group | Placebo | Rilonacept 160 mg | Open-Label Extension (OLE) Rilonacept 160 mg
Started | 0 (After week 24, all subjects are treated with Open label rilonacept.) | 0 | 101
Completed | 0 | 0 | 81
Not Completed | 0 | 0 | 20
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Death | 0 | 0 | 2
Not completed — Sponsor Decision | 0 | 0 | 15
Not completed — Pregnancy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Open-Label Rilonacept 160 mg: 57 new subjects entered the study directly into the OLE. This was not part of the double blind or randomized withdrawal portion of the results. The 44 subjects who completed Parts A and B were not included in this category for baseline characteristics. Pediatric subjects , age 7 or older, received rilonacept dosed 2.2 mg/kg weekly up to 160 mg during the OLE.
- Total: Total of all reporting groups
Arm/Group | Placebo | Rilonacept 160 mg | Open-Label Rilonacept 160 mg | Total
Number analyzed (Participants) | 24 | 23 | 57 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 8 | 8
  Between 18 and 65 years | 17 | 20 | 46 | 83
  >=65 years | 7 | 3 | 3 | 13
Age Continuous [Mean (Standard Deviation); unit: years] | 55.5 (14.7) | 45.9 (16) | 37.7 (17.2) | 43.6 (17.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 37 | 68
  Male | 8 | 8 | 20 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Everyone in Part A and Part B of the study was non hispanic and white.
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 24 | 23 | 56 | 103
    Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 24 | 23 | 57 | 104
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 23 | 57 | 104

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week-6 (Part A) Endpoint in Mean Key Symptom Score (KSS)
Description: The mean Key Symptom Score (KSS --from the validated, patient-administered Daily Health Assessment Form(DHAF)) was the average on a 0-10 scale (0=None, 10=Very Severe) of 5 separate scales -- rash, feeling of fever/chills, joint pain, eye redness/pain, and fatigue). KSS was averaged over two 21-day daily reporting periods (the 3 weeks prior to both baseline and week 6). In part A, a negative change in mean values indicated improvement under treatment with rilonacept in symptoms.
  The DHAF was used because it is a validated instrument to collect subject's self-reported responses.
Time Frame: Baseline (Days -21 to -1) and Week 6 (Days 21-42)
Population: Cryopyrin Associated Autoinflammatory Syndrome (CAPS) is a rare, orphan, hereditary disease. There are several hundred CAPS cases in the United States.
Measure: Mean (Standard Deviation); unit: Units of a Scale
Arm/Group | Placebo | Rilonacept 160 mg
Number analyzed (Participants) | 24 | 23
Units of a Scale
  Baseline Part A | 2.4 (1.5) | 3.1 (1.9)
  Endpoint Part A (Week 6) in KSS | 2.1 (1.6) | 0.5 (0.5)
  Change to Week 6 in KSS | -0.3 (0.7) | -2.6 (1.9)
Statistical Analysis 1: Comparison: Placebo vs Rilonacept 160 mg; The sample size calculations at the time suggested 50 subjects would be enrolled at baseline. The Full Analysis Set (FAS) was used. The FAS included subjects who received at least one dose of rilonacept. Last observation carried forward was used; Test type: Superiority or Other; p < .0001, ANCOVA; Comparison of p-value was a parametric ANCOVA main effects model with part A Baseline variable as covariate and treatment

2. Primary Outcome: Mean Change in Key Symptom Score (KSS) From Week 15 to Week 24 (During the Randomized Withdrawal Phase or Part B)
Description: The mean Key Symptom Score (KSS --from the validated, patient-administered DHAF) was the average on a 0-10 scale (0=None, 10=Very Severe) of 5 separate scales -- rash, feeling of fever/chills, joint pain, eye redness/pain, and fatigue).
  Subjects all received rilonacept 160 mg from week 6 through week 14. At week 15, subjects were re-randomized in a 1:1 ratio between Placebo and rilonacept 160 mg. Subjects baseline period was the 21-day period prior to week 15 randomization.
  A positive score indicated a worsening of symptoms versus an active treatment rilonacept baseline period.
Time Frame: Week 15 through Week 24 (randomized withdrawal)
Population: Subjects were re-randomized as part of the randomized withdrawal period (Part B). Subjects were not necessarily assigned the same treatment as in the first double-blind portion (Part A). Subjects were analyzed using last observation carried forward.
Measure: Mean (Standard Deviation); unit: Units of a Scale
Arm/Group | Placebo | Rilonacept 160 mg
Number analyzed (Participants) | 23 | 22
Units of a Scale
  Baseline Part B | 0.2 (0.4) | 0.3 (0.3)
  Endpoint Part B (Week 24) in KSS | 1.2 (1.0) | 0.4 (0.5)
  Change to Week 24 in KSS | 0.9 (0.9) | 0.1 (0.4)
Statistical Analysis 1: Comparison: Placebo vs Rilonacept 160 mg; Subjects received rilonacept 160 mg for 9 weeks (weeks 6-15), and then were re-randomized 1:1 into either Placebo or rilonacept 160 mg. The endpoint for the period was 9 weeks later (week 24). The sample size calculations at the time suggested 50 subjects would be enrolled at baseline. The Full Analysis Set (FAS) was used. The FAS included subjects who received at least one dose of rilonacept. Last observation carried forward was used; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]

3. Other Pre Specified Outcome: Mean Change From Baseline to Endpoint (Week 6) in Number of Disease Flare Days Per Patient
Description: A Disease flare day was any day where the mean Key Symptom Score (KSS) was greater than 3. The KSS was the average on a 0-10 scale (0=None, 10=Very Severe) of 5 separate scales -- rash, feeling of fever/chills, joint pain, eye redness/pain, and fatigue). KSS was calculated for 21 Day Periods at baseline and at the endpoint (from Weeks 3 - 6). The difference in the number of flares between the two periods was averaged for all subjects.
  The DHAF was used because it is a validated instrument to collect subject's self-reported responses. It was the basis for the KSS and the flare day count.
Time Frame: Baseline to Week 6 (Part A)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Rilonacept 160 mg
Number analyzed (Participants) | 24 | 23
Days
  Baseline Part A | 6.2 (6.0) | 8.6 (7.2)
  Endpoint Part A (Week 6) in Flare Days | 5.0 (6.1) | 0.1 (0.5)
  Change to Week 6 in Flare Days | -1.2 (3.6) | -8.4 (7.1)
Statistical Analysis 1: Comparison: Placebo vs Rilonacept 160 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]

4. Other Pre Specified Outcome: Change From Baseline to Endpoint (Week 6) in Physician's Global Assessment
Description: The Physician's Global Assessment was an evaluation at each visit on a scale of 0=no disease activity to 10=severe disease activity. A negative value in change in Physician's Global Assessment is indicative of an improvement.
Time Frame: Baseline to Week 6 (Part A)
Measure: Mean (Standard Deviation); unit: Units of a Scale
Arm/Group | Placebo | Rilonacept 160 mg
Number analyzed (Participants) | 24 | 23
Units of a Scale
  Baseline Part A | 4.7 (2.0) | 5.6 (1.7)
  Endpoint Part A in Physician's Global Assessment | 5.0 (2.5) | 1.5 (1.4)
  Change to Week 6 in Physician's Global Assessment | 0.2 (2.1) | -4.2 (2.4)
Statistical Analysis 1: Comparison: Placebo vs Rilonacept 160 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Comparison P-Value was a parametric ANCOVA main effects model with Part A Baseline variable as covariate and treatment

5. Other Pre Specified Outcome: Mean Change From Baseline to Endpoint (Week 6) in Patient's Global Assessment
Description: The Patient's Global Assessment was a question on the Daily Health Assessment Form "Considering all the ways that Familial Cold Autoinflmatory Syndrome (FCAS) /Muckle-Wells Syndrome (MWS) affects you, please rate how you are doing based on the following scale" 0=very well to 10=very poor. A negative value in change in Patient's Global Assessment is indicative of an improvement.
Time Frame: Baseline to Week 6 (Part A)
Measure: Mean (Standard Deviation); unit: Visual Analog Scale
Arm/Group | Placebo | Rilonacept 160 mg
Number analyzed (Participants) | 24 | 23
Visual Analog Scale
  Baseline in Part A | 3.1 (2.0) | 3.6 (2.1)
  Endpoint Part A in Patient's Global Assessment | 2.7 (1.8) | 0.9 (1.1)
  Change to Week 6 in Patient's Global Assessment | -0.4 (1.1) | -2.7 (2.2)
Statistical Analysis 1: Comparison: Placebo vs Rilonacept 160 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < .0001, ANCOVA; Comparison p-value is a parametric ANCOVA main effects model with Part A Baseline variable as covariate and treatment

6. Other Pre Specified Outcome: Median Change From Baseline to Week 6 (Part A) Endpoint in C-Reactive Protein (mg/L)
Description: An abnormal value for CRP was considered > 8.4 mg/L.
Time Frame: Baseline to Endpoint of Part A
Measure: Median (Standard Deviation); unit: Milligrams per Liter
Arm/Group | Placebo | Rilonacept 160 mg
Number analyzed (Participants) | 24 | 23
Milligrams per Liter
  Baseline Part A | 25.2 (15.7) | 20.1 (14.7)
  Endpoint Part A in CRP | 21.8 (23.9) | 1.3 (2.2)
  Change to Part A Endpoint in CRP | -2.1 (15.5) | -18.4 (14.3)
Statistical Analysis 1: Comparison: Placebo vs Rilonacept 160 mg; Please note that the changes are medians (not means). The sample size calculations at the time suggested 50 subjects would be enrolled at baseline. The Full Analysis Set (FAS) was used. The FAS included subjects who received at least one dose of rilonacept. Last observation carried forward was used; Test type: Superiority or Other; p < 0.0001, ANCOVA; Comparison p-value was a parametric ANCOVA main effects model with Part A Baseline variable as covariate and treatment

7. Other Pre Specified Outcome: Median Change From Baseline to Week 6 (Part A) Endpoint in Serum Amyloid A (mg/L)
Description: An abnormal value for SAA was considered > 6.4 mg/L.
Time Frame: Baseline to Endpoint of Part A
Measure: Median (Standard Deviation); unit: Milligrams per Liter
Arm/Group | Placebo | Rilonacept 160 mg
Number analyzed (Participants) | 24 | 23
Milligrams per Liter
  Baseline Part A | 63.5 (122.3) | 49.5 (48.3)
  Endpoint Part A in SAA | 39.7 (153.7) | 2.5 (4.0)
  Change to Endpoint in SAA | -2.8 (79.7) | -48.5 (48.5)
Statistical Analysis 1: Comparison: Placebo vs Rilonacept 160 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.01, ANCOVA; Comparison p-value was a parametric ANCOVA main effects model with Part A Baseline variable as covariate and treatment

8. Other Pre Specified Outcome: Number of Subjects With at Least 30% Improvement in Key Symptoms Scores (KSS) From Baseline to Endpoint (Week 6)
Description: The mean Key Symptom Score (KSS --from the validated, patient-administered Daily Health Assessment Form(DHAF)) was the average on a 0-10 scale (0=None, 10=Very Severe) of 5 separate scales -- rash, feeling of fever/chills, joint pain, eye redness/pain, and fatigue).
Time Frame: Baseline to Endpoint (Week 6)
Measure: Number; unit: Participants
Arm/Group | Placebo | Rilonacept 160 mg
Number analyzed (Participants) | 24 | 23
Participants | 7 | 22
Statistical Analysis 1: Comparison: Placebo vs Rilonacept 160 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Fisher Exact

9. Other Pre Specified Outcome: Number of Subjects With at Least 50% Improvement in Key Symptoms Scores (KSS) From Baseline to Endpoint (Week 6)
Description: as for outcome 8
Time Frame: Baseline to Week 6 (Part A)
Measure: Number; unit: Participants
Arm/Group | Placebo | Rilonacept 160 mg
Number analyzed (Participants) | 24 | 23
Participants | 2 | 20
Statistical Analysis 1: Comparison: Placebo vs Rilonacept 160 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Fisher Exact

10. Other Pre Specified Outcome: Number of Subjects With at Least 75% Improvement in Key Symptoms Scores (KSS) From Baseline to Endpoint (Week 6)
Description: as for outcome 8
Time Frame: Baseline to Week 6 (Part A)
Measure: Number; unit: Participants
Arm/Group | Placebo | Rilonacept 160 mg
Number analyzed (Participants) | 24 | 23
Participants | 0 | 16
Statistical Analysis 1: Comparison: Placebo vs Rilonacept 160 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Fisher Exact

11. Other Pre Specified Outcome: Summary of Mean Change From Baseline to Open-Label Extension Week 72 in KSS
Description: OLE Week 72 was the last timepoint at which efficacy was measured in the study. 56 of the 101 OLE subjects were included in the analysis.
  The mean Key Symptom Score (KSS --from the validated, patient-administered Daily Health Assessment Form(DHAF)) was the average on a 0-10 scale (0=None, 10=Very Severe) of 5 separate scales -- rash, feeling of fever/chills, joint pain, eye redness/pain, and fatigue).
  A negative change in mean values indicated improvement in symptoms.
Time Frame: From Baseline (week 0) to OLE Week 72
Population: 44 subjects entered from part A of the study, and 12 subjects entered directly into the OLE. No placebo subjects were in the OLE.
Measure: Mean (Standard Deviation); unit: Units of a scale
Arm/Group | Rilonacept 160 mg
Number analyzed (Participants) | 56
Units of a scale
  Baseline | 2.6 (1.6)
  Endpoint (OLE Week 72) in KSS | 0.4 (0.5)
  Change to Endpoint (OLE Week 72) in KSS | -2.3 (1.6)

12. Other Pre Specified Outcome: Change From Baseline to Open-Label Extension Week 72 in Patient's Global Assessment
Description: The Patient's Global Assessment was a question on the Daily Health Assessment Form "Considering all the ways that FCAS/MWS affects you, please rate how you are doing based on the following scale" 0=very well to 10=very poor. A negative value in change in Patient's Global Assessment is indicative of an improvement.
  OLE Week 72 was the last timepoint at which efficacy was measured in the study. 56 of the 101 OLE subjects were included in the analysis.
Time Frame: From Baseline (Week 0) to OLE Week 72
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units of a Scale
Arm/Group | Rilonacept 160 mg
Number analyzed (Participants) | 56
Units of a Scale
  Baseline | 3.4 (1.9)
  OLE Week 72 in Patient's Global Assessment | 0.4 (0.6)
  Change to OLE Wk 72 in Patient's Global Assessment | -3.0 (2.0)

13. Other Pre Specified Outcome: Change From Baseline to Open-Label Extension Week 72 in Number of Disease Flare Days
Description: OLE Week 72 was the last timepoint at which efficacy was measured in the study. 56 of the 101 OLE subjects were included in the analysis.
  A Disease flare day was any day where the mean Key Symptom Score (KSS) was greater than 3. The mean Key Symptom Score (KSS --from the validated, patient-administered Daily Health Assessment Form(DHAF)) was the average on a 0-10 scale (0=None, 10=Very Severe) of 5 separate scales -- rash, feeling of fever/chills, joint pain, eye redness/pain, and fatigue).
Time Frame: From Baseline (Week 0) to OLE Week 72
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | Rilonacept 160 mg
Number analyzed (Participants) | 56
Number of Days
  Baseline | 7.3 (6.4)
  Endpoint in OLE Week 72 Disease Flare Days | 0.6 (3.0)
  Change to OLE Week 72 in Disease Flare Days | -6.7 (6.9)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) were reported for all phases (double blind, randomized withdrawal, and OLE) of the study. There were no SAEs for subjects on placebo during Parts A or B. Other adverse events were shown for the six week double-blind period.
Description: All serious adverse events were considered not related to receiving rilonacept by the physician at the site. Other adverse events were shown if a minimum of 2 subjects (approximately 4 percent of the Part A subjects) had the event during the 6-week, double-blind period.
Arm/Group | Rilonacept 160 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 7/104 | 0/24
Other Adverse Events (participants affected / at risk) | 17/23 | 13/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rilonacept 160 mg (N=104) | Placebo (N=24)
Meningitis pneumococcal (Infections and infestations) | 1 (1) | 0 — This SAE resulted in subject's death. The investigator reported that this was not drug-related. Interleukin-1 blockade may interfere with immune response to infections. Life-threatening infections have been reported in patients taking rilonacept.
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 — Treatment Emergent Serious Adverse Events are reported for all phases of the study.
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Sciatica (Nervous system disorders) | 1 (1) | 0 — Sciatica was the only serious adverse event during the first 24 weeks of the study. It occurred during the single-blind period between Parts A and B when all subjects received rilonacept.
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0
Renal Colic (Renal and urinary disorders) | 1 (1) | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0
Arteriosclerosis of the coronary artery (Cardiac disorders) | 1 (1) | 0 — The arteriosclerosis of the coronary artery resulted in the subject's death. The investigator reported that this was deemed not to be drug-related but related to the patient's underlying history of CHD.
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rilonacept 160 mg (N=23) | Placebo (N=24)
Injection Site Reaction (General disorders) | 11 | 3 — Included erythema, pruritis, swelling, bruising, inflammation, mass, or pain at the injection site. All injection site reactions in part a were mild or moderate in severity.
Sinusitis (Infections and infestations) | 2 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 6 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 1 | 3
Abdominal pain, upper abdomen (Gastrointestinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoesthesia (Nervous system disorders) | 2 | 0
Stomach Discomfort (Gastrointestinal disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
Cryopyrin Associated Periodic Syndrome (CAPS) is a rare disease with only a few hundred cases in the US.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI,after completion of a trial,is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review;provided that the sponsor can remove confidential or proprietary information from such communications. The sponsor cannot require other changes to the communication and cannot extend the embargo.